CLINICAL TRIAL: NCT04152447
Title: Virtual Reality for Pain Management in Orthopaedic Patients: A Prospective Randomized Control Pilot Study
Brief Title: Virtual Reality for Pain Management in Orthopaedic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Principal Investigator, Marilyn Heng, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018P002763
Record Dates: First submitted 2019-10-16; First posted 2019-11-05 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Pain, Musculoskeletal
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of care (No Intervention): This arm describes the standard protocol used to aid in orthopedic recovery.
- VR device (Active Comparator): Patients randomly assigned to the experimental arm of the study were provided an Oculus Go™ device for the duration of their hospitalization. The device featured a headset with a 1280 x 1440, 60 Hz refresh rate LCD display, spatial audio (via built-in speakers; headphones were not provided or used to our knowledge, despite compatibility) and the ability to track 3 degrees of rotational freedom; it was compatible with glasses and included a soft, adjustable strap for optimal, user-based fit. A single controller, capable of recognizing hand motion, pointing, and clicking was also included.
  Interventions: Device: VR device

INTERVENTIONS:
Device: VR device — Patients use a VR device
  Arms: VR device

SUMMARY:
1. Investigators will determine the feasibility of a virtual reality pain control program (VR-PCP) as a non-pharmacologic adjunct for pain management while in the hospital (i.e. patient ability and willingness to use the system measured by average time spent on the device).
2. Investigators will evaluate if there is a difference between the average daily use of opioid medications taken by patients who received usual care pain management versus patients using a VR-PCP.
3. Investigators will assess for differences in short-term postoperative patient-reported pain intensity (PROMIS Patient Intensity v1.0) for patients who received usual care pain management versus those who also have access to a VR-PCP.

DETAILED DESCRIPTION:
Orthopedic surgeons rank third amongst physician prescribers of opioids to adults in the United States4. The deleterious effects of the opioid epidemic have been well studied at both the individual and population level.2 3 Orthopaedic trauma patients in particular have high rates of psychological stress and disability related to protracted narcotic usage 5. However, opioid medications may not need to be the mainstay of pharmacologic pain management for patients with orthopaedic injuries. For example, one recent study from the Netherlands showed that 82% of patients with ankle fractures treated in the United States were prescribed opioids at discharge, whereas only 6% of Dutch patients were given narcotics. 6

Non-pharmacologic interventions for pain management in the acute orthopaedic injury setting deserve full investigation. Virtual reality for pain management has been used in burn patients, pediatric patients, for procedures under local anesthesia and in the chronic pain setting. Results of these investigations are promising and demonstrate reduced narcotic usage and improved pain scores.7 8 9 Currently, there are no published reports on the use of virtual reality for pain management in the orthopaedic literature. By investigating VR as a non-pharmacologic intervention for pain, orthopaedic trauma patients may be able to avoid the known risks of narcotic medication while still controlling their pain and regaining function after their injury. Our study will lay groundwork for longer-term studies to evaluate the impact of virtual reality on functional outcomes, opioid usage after hospital discharge and patient satisfaction scores. VR can also be investigated for post-operative pain control across other orthopedic subspecialties.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Patients who sustained factures treated with open reduction internal fixation. Polytrauma patients whose fractures are definitively fixed in one discrete operating room visit will be included.

Exclusion Criteria:

* Cognitive impairment
* Injuries requiring staged surgical fixation (i.e. ex-fix to ORIF)
* Seizure disorder or other contraindication to VR usage
* Significant medical complications during hospitalization precluding use of a VR headset
* Significant surgical complication during hospitalization requiring unanticipated return to the operating room during index admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Heng, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: The standard of care for orthopaedic trauma patients is a multimodal pain management approach aimed at minimizing narcotic usage, particularly in our geriatric fracture patients. Standard practice is to never give so much opioids, to any patient, that the renders them confused or obtunded. In this study, we follow MGH nursing protocols for the group receiving the standard of care.
Period: Overall Study
Arm/Group | Standard of Care | VR Device
Started | 16 | 19
Completed | 13 | 14
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Treatment plan switched to an ineligible criteria | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Found ineligible after enrolling | 1 | 1
Not completed — Did not receive VR headset in time. | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: The usual care for pain management at our institution consists of standing Tylenol, oxycodone PRN and IV Dilaudid PRN for breakthrough pain. Existing MGH nursing protocols evaluate when to give PRN narcotics to patients based on functional pain levels and are aimed at minimizing narcotic use. In elderly patients, the PRN dose of narcotics prescribed is generally half that of their younger counterparts (2.5-5mg q4h PRN versus 5-10mg q4h PRN in younger patients).
  Geriatric fracture patients admitted to the orthopaedic trauma service are comanaged with geriatricians who also carefully monitor the effects of these medications. In this manner, the standard of care for orthopaedic trauma patients is a multimodal pain management approach aimed at minimizing narcotic usage, particularly in our geriatric fracture patients. Standard practice is to never give so much opioids, to any patient, that the renders them confused or obtunded.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | VR Device | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 7 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 3 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Opioid Usage During the Postoperative Hospitalization
Description: Opioid usage during the postoperative hospitalization measured in average daily morphine milligram equivalents (MME). Higher number is a worse outcome.
Time Frame: Post-operative period, an average of 3 days
Population: This population involves the eligible patient population that has received opioids following surgery.
Measure: Mean (95% Confidence Interval); unit: Morphine milligram equivalents (MME)/day
Arm/Group | Standard of Care | VR Device
Number analyzed (Participants) | 13 | 14
Morphine milligram equivalents (MME)/day | 30.3 [12.7 to 42.2] | 30.8 [18.7 to 47.2]

2. Secondary Outcome: Length of Stay
Description: Length of Stay is measured as days following surgery and before discharge.
Time Frame: Post-operative period, an average of 3 days
Population: The population is the population enrolled in the study: patients 18 or over who are opioid naïve and have had surgery.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Standard of Care | VR Device
Number analyzed (Participants) | 13 | 14
days | 2.5 [2 to 4] | 2 [1 to 4]

3. Secondary Outcome: Patient-reported Pain Scores
Description: Patients had to answer a series of questionnaires regarding their pain level at baseline, and daily during hospitalization. The scores were tallied up. This scale is referred to as the PROMIS Pain Intensity Scale v1.0, which tracks patient reported outcomes on a scale where 3 is the minimum and 15 is the maximum. PROMIS scores are taken daily post-operation, and the score reported is the reflection of the average PROMIS score of the post-operative days, since patients did not stay for the same length following surgery. Higher score is a worse outcome. Minimum value is 0, Maximum value is 100.
Time Frame: Post-operative period, an average of 3 days
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard of Care | VR Device
Number analyzed (Participants) | 13 | 14
score on a scale | 9.62 [9.0 to 11.3] | 9.0 [7.0 to 11.5]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the span of 1 year and 2 months, from the consent of the first patient through the discharge of the final patient from the hospital. For each patient, Adverse events were tracked on the period from baseline to discharge from the hospital, which differed per patient but averaged to around 3 days following surgery.
Description: Given the non-invasive nature of the VR headsets, we subcategorize serious Adverse Events as device-related or non device-related. For non-medical issues, we handled them on an event-to-event basis, informing the study staff and triaging. When postoperative complications occur in a patient enrolled in the study, the PI will immediately be notified. The PI will be responsible for collecting laboratory data and medical history to ensure that the AE was not device related.
Arm/Group | Standard of Care | VR Device
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT04152447/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT04152447/SAP_002.pdf